CLINICAL TRIAL: NCT01552681
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial of Baminercept, a Lymphotoxin-beta Receptor Fusion Protein, for the Treatment of Primary Sjögren's Syndrome (ASJ02)
Brief Title: Baminercept, a Lymphotoxin-Beta Receptor Fusion Protein, for Treatment of Sjögren's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Expired experimental study agent, no additional supply available.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ASJ02
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2018-12

CONDITIONS: Primary Sjögren's Syndrome
Keywords: baminercept treatment
MeSH Terms: interventions — baminercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baminercept (Experimental): Subcutaneous injections of 100 mg every week for 24 weeks
  Interventions: Biological: Baminercept
- Placebo (Placebo Comparator): Subcutaneous injections of matched placebo every week for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Baminercept — Subjects randomized to baminercept (2:1) will receive 24 weekly injections of 100 mg administered subcutaneously starting at the Day 0 visit and ending at Week 23.
  Other Names: lymphotoxin-beta receptor-immunoglobulin fusion protein
  Arms: Baminercept
Other: Placebo — Subjects randomized to placebo will receive 24 weekly injections of 100 mg administered subcutaneously starting at the Day 0 visit and ending at Week 23.
  Other Names: baminercept placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to find out if the experimental study agent, baminercept, is effective in treating patients with Sjögren's syndrome. The study will also determine if the study agent can be safely given to patients with Sjögren's syndrome; examine how it affects symptoms of the disease; and attempt to understand how baminercept affects the underlying mechanisms of Sjögren's syndrome and the immune system.

DETAILED DESCRIPTION:
Sjögren's syndrome is an autoimmune disorder in which a person's own immune cells attack the body's tear and salivary glands. This disease is the second most common autoimmune disorder, affects close to four million people in the U.S., and has no known cause. About one-third of patients with Sjögren's syndrome have enlarged parotid glands (the largest salivary glands, the glands that make saliva); inflammation of organs such as the lungs and joints may also occur. There is no known effective treatment other than measures that can relieve symptoms. One of the most bothersome symptoms is dryness of the eyes and mouth. Eye drops and saliva stimulants (which help make more saliva) are common treatments. When other organs are affected, symptoms are treated with corticosteroids (prednisone), non-steroidal anti-inflammatory drugs (NSAIDs, such as ibuprofen and naproxen), hydroxychloroquine (Plaquenil®) or other medications that suppress the immune system. These drugs may curb or kill cells of the immune system, but they are not always helpful, do not cure Sjögren's syndrome, and can have many side effects.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent;
* Between the ages of 18-75 years (inclusive);
* Body weight ≥ 40 kg;
* Meets the revised European criteria proposed by the American-European Consensus Group for primary Sjögren's Syndrome at screening. These criteria include 3 of the following 4 items:

  * ocular symptoms;
  * oral symptoms;
  * Schirmer's I test showing less than 6 mm of wetting per five minutes in at least one eye, or filamentary keratitis on slit lamp examination, or positive lissamine green staining; or
  * diminished salivary production (unstimulated whole salivary flow rate ≤ 1.5 mL/15 min); PLUS, either:
  * a positive test for serum SS-A and/or SS-B antibodies, or
  * focal lymphocytic sialadenitis, with a focus score ≥ 1.0 per 4 millimeters ^2(mm^2) on minor salivary biopsy.
* Stimulated salivary flow of ≥ 0.1 mL/minute (min) (at screening);
* Has one or more of the following systemic manifestations of Sjögren's Syndrome that are not life-threatening:

  * fatigue (as measured by > 50 mm on a 100 mm VAS);
  * joint pain (as measured by > 50 mm on a 100 mm VAS);
  * peripheral neuropathy (documented by nerve conduction velocity study);
  * interstitial lung disease (documented by radiography and/or altered pulmonary function tests;
  * leukocytoclastic vasculitis;
  * renal tubular acidosis;
  * interstitial nephritis;
  * severe parotid swelling;
  * other extraglandular manifestations causing organ system dysfunction.
* If taking prednisone (or equivalent corticosteroid), the dose must be ≤ 10 mg/day and stable for at least 4 weeks prior to Screening;
* If taking hydroxychloroquine, the dose must be stable for at least 12 weeks prior to Screening;
* If taking a cholinergic stimulant (e.g. pilocarpine, cevimeline), the dose must be stable for at least 4 weeks prior to Screening;
* Subjects must agree not to become pregnant or to impregnate a female. Because of the risk involved, participants and their partners (if of reproductive potential) must use two methods of birth control. They must continue to use both methods until 6 months after stopping study drug. Two of the birth control methods listed below may be chosen:

  * Hormonal contraception;
  * Male or female condoms with or without spermicide;
  * Diaphragm or cervical cap with a spermicide;
  * Intrauterine device (IUD).

Exclusion Criteria:

* Has an active infection excluding superficial cutaneous fungal or viral infections;
* Has a chronic or persistent infection that might be worsened by immunosuppressive treatment (e.g., human immunodeficiency virus [HIV], hepatitis B, hepatitis C, or tuberculosis);
* History of TB or positive intradermal skin test for purified protein derivative (PPD); positive Mantoux test defined as 10 mm of induration (size of raised bump, not redness), or equivalent positive TB test result, as per country clinical standards, during the screening period. Subjects whose PPD induration is ≥ 5 mm but < 10 mm are eligible for the study if they had a negative chest x-ray during the screening period. There must be no other clinical evidence of TB on physical examination of the subject. Note: Subjects who have had prior adequate prophylaxis treatment for latent TB with an appropriate course of isoniazid or equivalent, per country standards, are not excluded from study participation. PPD should not be administered within 6 weeks of a live-virus vaccine;
* History of recurrent significant infections or occurrence of a serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within twelve weeks prior to Day 0;
* Receipt of live vaccine within six weeks prior to Day 0;
* History or presence of primary or secondary immunodeficiency;
* History of any life-threatening allergic reactions;
* Is a pregnant or nursing female;
* Ongoing anticoagulant therapy, which is a contraindication for labial salivary biopsy or tonsil biopsy;
* Concurrent use of anticholinergic agents, such as tricyclic antidepressants, antihistamines, phenothiazines, antiparkinsonian drugs, anti-asthmatic medications, or gastrointestinal (GI) medications that cause xerostomia in more than 10% of patients;
* Treatment with any of the following within the defined period prior to Screening:

  * 2 years for rituximab;
  * 24 weeks for cyclophosphamide;
  * 8 weeks for azathioprine, cyclosporine, methotrexate, or mycophenolate mofetil;
  * 4 weeks for intravenous immunoglobulin;
  * 4 weeks for etanercept;
  * 8 weeks for adalimumab;
  * 12 weeks for infliximab.
* Prednisone (or equivalent corticosteroid) > 10 mg/day;
* A definite diagnosis of RA, SLE, systemic sclerosis, or dermatomyositis;
* A history of alcohol or substance abuse within 12 months of the screening visit;
* A history of head and neck radiation therapy, sarcoidosis, or graft-versus-host disease;
* A history of malignancy, except for a resected basal or major squamous cell carcinoma, cervical dysplasia, or in situ cervical cancer Grade I, within the last five years;
* Severe pulmonary disease as manifested by one of the following at Screening:

  * Resting oxygen saturation < 92%;
  * Force vital capacity (FVC) < 50% predicted;
  * Diffusion lung capacity for carbon monoxide (DLCO) < 50%;
* Abnormal laboratory results for the following parameters at the screening visit:

  * Absolute neutrophil count (ANC): < 1,500/mm^3;
  * Platelets: < 100,000/mm^3;
  * Hemoglobin: < 9 grams (g)/deciliter (dL);
  * Serum creatinine: ≥ 2.0 mg/dL;
  * AST: > 1.5x upper limit of normal, or
  * ALT: > 1.5x upper limit of normal.
* A psychiatric disorder rendering the subject incapable of providing informed consent;
* Plans for foreign travel to countries other than Canada or Western Europe within the treatment period;
* Inability or unwillingness to follow the protocol;
* Any condition or treatment that, in the opinion of the investigator, places the subject at an unacceptable risk as a participant in the trial;
* Rochester substudy subjects who meet the following criteria are disqualified from enrolling in the tonsil biopsy substudy if they:

  * Have any side effects to local anesthetics (e.g., lidocaine);
  * Have any side effects to silver nitrate;
  * Do not have tonsils;
  * Are not able to go 48 hours without any NSAIDS;
  * Are not able to go 2 weeks without acetylsalicylic acid (aspirin).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. William St. Clair, MD, Study Chair — Duke University; Judith A. James, MD, Study Chair — Oklahoma Medical Research Foundation
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools that are available to researchers who register online and subsequently receive DAIT approval.

REFERENCES:
- [Result] St Clair EW, Baer AN, Wei C, Noaiseh G, Parke A, Coca A, Utset TO, Genovese MC, Wallace DJ, McNamara J, Boyle K, Keyes-Elstein L, Browning JL, Franchimont N, Smith K, Guthridge JM, Sanz I, James JA; Autoimmunity Centers of Excellence. Clinical Efficacy and Safety of Baminercept, a Lymphotoxin beta Receptor Fusion Protein, in Primary Sjogren's Syndrome: Results From a Phase II Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Rheumatol. 2018 Sep;70(9):1470-1480. doi: 10.1002/art.40513. Epub 2018 Jul 18. PMID 29604186
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/pages/default.aspx?wt.ac=tnHome
- Available data/document: Study Protocol: SDY823 — http://www.immport.org/immport-open/public/home/home — ImmPort study identifier is SDY823.
- Available data/document: Complete set of descriptive data and results: SDY823 — http://www.immport.org/immport-open/public/home/home — ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. This archive is in support of the NIH mission to share data with the public.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from nine sites in the United States. The first site was activated in July 2012 and the last participant was randomized on 22 July 2014.
Groups:
- Baminercept 100 mg: Participants were randomized to receive one subcutaneous injection of 100 mg baminercept every week for 24 weeks.
- Placebo: Participants were randomized to receive one subcutaneous injection of placebo every week for 24 weeks.
Period: Overall Study
Arm/Group | Baminercept 100 mg | Placebo
Started | 33 | 19
Completed | 28 | 18
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Subject moved away | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat population included all randomized subjects who received at least one dose of either baminercept or placebo and had a screening stimulated salivary flow assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Baminercept 100 mg | Placebo | Total
Number analyzed (Participants) | 33 | 19 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.9) | 54.7 (11.0) | 52.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 18 | 49
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 29 | 17 | 46
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 28 | 16 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 19 | 52
Body Weight [Mean (Standard Deviation); unit: kg] — Body weight at the baseline visit. Weight of 40 kg or greater was required to enter the study.
  kg | 75.5 (20.4) | 79.2 (19.3) | 76.9 (19.9)
Height [Mean (Standard Deviation); unit: cm] — Height at the baseline visit. Data were not available for six participants who received baminercept and four participants who received placebo.
  cm | 164.4 (7.1) | 163.2 (7.7) | 164.0 (7.3)
Stimulated Salivary Flow Rate [Mean (Standard Deviation); unit: mL/min] — After an unstimulated salivary flow assessment the participant was administered a single 5-mg dose of pilocarpine to stimulate saliva production. One hour after the administration of pilocarpine the participant spit into a preweighed 50-cm centrifuge tube for 15 minutes. The sample was weighed to determine the volume (1 g = 1 mL) of saliva. The volume of saliva (mL) was divided by the duration of the test (minutes) to calculate the stimulated salivary flow rate (mL/min). A stimulated salivary flow rate of ≥ 0.1 mL/min (min) was required to enter the study.
  mL/min | 0.4 (0.5) | 0.5 (0.3) | 0.5 (0.4)
European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) Score [Mean (Standard Deviation); unit: units on a scale] — The ESSDAI is a clinical index that measures Sjogren's syndrome disease activity. A physician scores the disease activity level of twelve organ-specific domains in 3 or 4 levels according to their severity. For example, for no disease activity the domain score equals 0 and for high disease activity the domain score equals 3 or 4. Each domain is assigned a weight between 1 and 6, and the domain score is multiplied by the domain weight. The sum of the weighted domain scores is the overall score, which can range from 0 to 123. A higher score indicates more disease activity.
  units on a scale | 2.7 (2.8) | 3.8 (4.2) | 3.1 (3.4)
Tender Joint Count [Mean (Standard Deviation); unit: units on a scale] — Tender Joint Count (TJC) is the number of tender joints based on the tenderness response of 28 joints examined. TJC possible values range from 0 to 28.
  units on a scale | 1.1 (2.0) | 5.0 (7.5) | 2.5 (5.1)
Swollen Joint Count [Mean (Standard Deviation); unit: units on a scale] — Swollen Joint Count (SJC) is the number of swollen joints based on swelling response of 28 joints examined. SJC possible values range from 0 to 28.
  units on a scale | 0.1 (0.5) | 0.2 (0.7) | 0.2 (0.6)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The physician's response to the question "Overall, how would you rate the Sjogren's Syndrome symptom activity of the subject?" A vertical mark on a 100 mm horizontal line rated 0 (Not active) to 100 (Very active). The range: 0 to 100, with 100 indicating severe symptoms.
  mm | 48.6 (20.6) | 50.3 (20.5) | 49.2 (20.4)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — A self-reported measure of perceived disease activity obtained by responding to the question "Overall, how would you rate your Sjogren's Syndrome symptom activity?" A vertical mark on a 100 mm line rated 0 (Not active) to 100 (Very active) determines the score. The range: 0 to 100, with 100 indicating severe symptoms.
  mm | 70.3 (16.5) | 73.5 (16.4) | 71.5 (16.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Screening in Stimulated Whole Salivary Flow at Week 24
Description: After an unstimulated salivary flow assessment the participant was administered a single 5-mg dose of pilocarpine to stimulate saliva production. One hour after the administration of pilocarpine the participant spit into a preweighed 50-cm centrifuge tube for 15 minutes. The sample was weighed to determine the volume (1 g = 1 mL) of saliva. The volume of saliva (mL) was divided by the duration of the test (minutes) to calculate the stimulated salivary flow rate (mL/min). Change from screening was computed as the value at Week 24 minus the screening value. A positive value in change from screening indicates an improvement and a negative value indicates worsening.
Time Frame: Screening to Week 24
Population: The Modified Intent-to-Treat population included all randomized subjects who received at least one dose of either baminercept or placebo with screening and post-screening stimulated salivary flow results. Participants missing Week 24 assessment were imputed from last post-screening assessment. Salivary flow results unavailable for one subject.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 32 | 19
mL/min | 0.0 (0.3) | 0.1 (0.2)
Statistical Analysis 1: Comparison: Baminercept 100 mg vs Placebo; Missing Week 24 assessments were imputed by carrying forward the last observed post-baseline value; Test type: Superiority or Other; p = 0.33, ANCOVA — P-value is testing for treatment effect using an analysis of covariance with adjustments for screening stimulated salivary flow

2. Secondary Outcome: Change From Screening in Stimulated Whole Salivary Flow at Week 48
Description: After an unstimulated salivary flow assessment the participant was administered a single 5-mg dose of pilocarpine to stimulate saliva production. One hour after the administration of pilocarpine the participant spit into a preweighed 50-cm centrifuge tube for 15 minutes. The sample was weighed to determine the volume (1 g = 1 mL) of saliva. The volume of saliva (mL) was divided by the duration of the test (minutes) to calculate the stimulated salivary flow rate (mL/min). Change from screening was computed as the value at Week 48 minus the screening value. A positive value in change from screening indicates an improvement and a negative value indicates worsening.
Time Frame: Screening to Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received >=1 dose of either baminercept or placebo and who had stimulated salivary flow results at screening and Week 48. Wk 48 stimulated salivary flow results were not available for N=7 subjects (e.g., N=6 in baminercept and N=1 in placebo group).
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 27 | 18
mL/min | 0.0 (0.3) | -0.1 (0.2)

3. Secondary Outcome: Change From Screening in Unstimulated Whole Salivary Flow at Week 24
Description: The participant spit into a preweighed 50-cm centrifuge tube for 15 minutes. The sample was weighed to determine the volume (1 g = 1 mL) of saliva. The volume of saliva (mL) was divided by the duration of the test (minutes) to calculate the unstimulated salivary flow rate (mL/min). Cholinergic stimulants such as pilocarpine or cevimeline were discontinued for 48 hours prior to the assessment and nothing was taken by mouth for 60 minutes or longer before or during saliva collection. Change from screening was computed as the value at Week 24 minus the screening value. A positive value in change from screening indicates an improvement and a negative value indicates worsening.
Time Frame: Screening to Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received >=1 dose of either baminercept or placebo and who had an unstimulated salivary flow assessment at screening and week 24. Data were not available for N=7 subjects (e.g., N=5 in baminercept and N=2 in placebo group).
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 28 | 17
mL/min | 0.1 (0.2) | 0.1 (0.1)

4. Secondary Outcome: Change From Screening in Unstimulated Whole Salivary Flow at Week 48
Description: The participant spit into a preweighed 50-cm centrifuge tube for 15 minutes. The sample was weighed to determine the volume (1 g = 1 mL) of saliva. The volume of saliva (mL) was divided by the duration of the test (minutes) to calculate the unstimulated salivary flow rate (mL/min). Cholinergic stimulants such as pilocarpine or cevimeline were discontinued for 48 hours prior to the assessment and nothing was taken by mouth for 60 minutes or longer before or during saliva collection. Change from screening was computed as the value at Week 48 minus the screening value. A positive value in change from screening indicates an improvement and a negative value indicates worsening.
Time Frame: Screening to Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had unstimulated salivary flow results at Screening and Week 48. Data were not available for six participants who received baminercept and one participant who received placebo.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 27 | 18
mL/min | 0.1 (0.1) | 0.1 (0.1)

5. Secondary Outcome: Change From Baseline in European League Against Rheumatism (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) at Week 24
Description: The ESSDAI is a clinical index that measures Sjogren's syndrome disease activity. A physician scores the disease activity level of twelve organ-specific domains in 3 or 4 levels according to their severity. For example, for no disease activity the domain score equals 0 and for high disease activity the domain score equals 3 or 4. Each domain is assigned a weight between 1 and 6, and the domain score is multiplied by the domain weight. The sum of the weighted domain scores is the overall score, which can range from 0 to 123. A higher score indicates more disease activity. Change from baseline was computed as the value at Week 24 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Baseline to Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had an ESSDAI score at Baseline and Week 24. Data were not available for five participants who received baminercept and two participants who received placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 28 | 17
units on a scale | -1.1 (2.3) | -0.4 (3.1)

6. Secondary Outcome: Percent of Subjects Classified as Responders According to the Patient Self-Assessment of Fatigue, Overall Dryness, and Joint Pain at Week 24
Description: Response is defined by 30% or more improvement (decrease) from baseline to week 24 in at least two of the three Visual Analog Scale (VAS) scores for patient self-assessment of symptoms of overall dryness, fatigue, and joint pain. On a 100-mm horizontal line the participant places a vertical mark to indicate a response. The range is 0 to 100, with 100 as the highest perceived overall fatigue, overall dryness, or joint pain.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had VAS results at Baseline and Week 24. Data were not available for four participants who received baminercept and one participant who received placebo.
Measure: Number; unit: Percent of participants
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 29 | 18
Percent of participants | 20.7 | 22.2

7. Secondary Outcome: Percent of Subjects Classified as Responders According to the Patient Self-Assessment of Fatigue, Overall Dryness, and Joint Pain at Week 48
Description: Response is defined by 30% or more improvement (decrease) from baseline to week 48 in at least two of the three Visual Analog Scale (VAS) scores for patient self-assessment of symptoms of overall dryness, fatigue, and joint pain. On a 100-mm horizontal line the participant places a vertical mark to indicate a response. The range is 0 to 100, with 100 as the highest perceived overall fatigue, overall dryness, or joint pain.
Time Frame: Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had VAS results at Baseline and Week 48. Data were not available for five participants who received baminercept and one participant who received placebo.
Measure: Number; unit: Percent of participants
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 28 | 18
Percent of participants | 21.4 | 5.6

8. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Scores for Sjogren's Syndrome Symptom Survey at Week 24
Description: On a 100-mm horizontal line the participant places a vertical mark to indicate responses to 14 questions about salivary and ophthalmic function. The range is 0 to 100, with 100 as the highest perceived difficulty, dryness, discomfort, swelling, thirst, dryness, severity, or sensitivity. Change from baseline was computed as the value at Week 24 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had VAS results at Baseline and Week 24. Data were not available for four participants who received baminercept and two participants who received placebo.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 29 | 17
mm
  Difficulty speaking due to dryness | -0.7 (29.1) | -9.2 (18.6)
  Difficulty swallowing due to dryness | -6.5 (23.6) | -10.1 (20.5)
  Dryness of mouth | -11.4 (27.2) | -12.7 (23.1)
  Dryness of throat | -4.9 (26.2) | -7.9 (25.7)
  Dryness of lips | -9.4 (24.7) | -10.8 (27.7)
  Dryness of tongue | -7.8 (25.5) | -8.9 (25.9)
  Thirst | -9.2 (29.4) | -11.9 (22.3)
  Oral discomfort in mouth | -4.4 (30.3) | -8.9 (23.0)
  Facial swelling | 0.3 (22.6) | 4.9 (18.1)
  Dry eye sensation | -1.6 (30.1) | -10.4 (25.0)
  Severity of sandy/gritty eye | -0.5 (37.4) | -7.3 (24.8)
  Blurry vision | -1.5 (35.6) | -7.6 (26.6)
  Sensitivity to bright lights | -6.6 (29.0) | -9.3 (16.4)
  Ease with which eyes feel tired | -7.6 (30.1) | -6.6 (16.9)

9. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Scores for Sjogren's Syndrome Symptom Survey at Week 48
Description: On a 100-mm horizontal line the participant places a vertical mark to indicate responses to 14 questions about salivary and ophthalmic function. The range is 0 to 100, with 100 as the highest perceived difficulty, dryness, discomfort, swelling, thirst, dryness, severity, or sensitivity. Change from baseline was computed as the value at Week 48 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had VAS scores at Baseline and Week 48. Data were not available for five participants who received baminercept and one participant who received placebo.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 28 | 18
mm
  Difficulty speaking due to dryness | -2.6 (33.4) | -2.8 (22.4)
  Difficulty swallowing due to dryness | -7.4 (24.8) | -1.3 (23.4)
  Dryness of mouth | -11.0 (24.1) | -6.6 (17.9)
  Dryness of throat | -4.0 (25.8) | -1.5 (20.9)
  Dryness of lips | -8.0 (21.3) | -3.4 (24.9)
  Dryness of tongue | -4.2 (22.2) | 1.3 (26.4)
  Thirst | -11.6 (25.8) | -5.8 (20.1)
  Oral discomfort in mouth | -9.6 (24.7) | 2.8 (22.4)
  Facial swelling | -3.7 (18.4) | 8.5 (24.4)
  Dry eye sensation | 0.5 (28.9) | -2.2 (21.2)
  Severity of sandy/gritty eye | 1.6 (39.2) | 4.3 (18.4)
  Blurry vision | -11.2 (35.8) | 5.1 (27.5)
  Sensitivity to bright lights | -10.2 (23.8) | -0.9 (22.5)
  Ease with which eyes feel tired | -11.3 (24.4) | -1.0 (22.7)

10. Secondary Outcome: Change From Baseline in Patient Self-Assessment of Fatigue, Overall Dryness, and Joint Pain at Week 24
Description: Three Visual Analog Scale (VAS) scores for patient self-assessment of symptoms of overall dryness, fatigue, and joint pain. On a 100-mm horizontal line the participant places a vertical mark to indicate responses to 3 questions. The range is 0 to 100, with 100 as the highest perceived tiredness, dryness, or joint pain. Change from baseline was computed as the value at Week 24 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had VAS scores at Baseline and Week 24. Data were not available for four participants who received baminercept and two participants who received placebo.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 29 | 17
mm
  Overall dryness | -8.3 (25.8) | -9.8 (21.6)
  Overall fatigue | -9.1 (26.9) | -9.3 (26.7)
  Degree of joint pain | -4.9 (25.6) | -8.7 (25.9)

11. Secondary Outcome: Change From Baseline in Patient Self-Assessment of Fatigue, Overall Dryness, and Joint Pain at Week 48
Description: Three Visual Analog Scale (VAS) scores for patient self-assessment of symptoms of overall dryness, fatigue, and joint pain. On a 100-mm horizontal line the participant places a vertical mark to indicate responses to 3 questions. The range is 0 to 100, with 100 as the highest perceived tiredness, dryness, or joint pain. Change from baseline was computed as the value at Week 48 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 28 | 18
mm
  Overall dryness | -10.8 (26.8) | -1.6 (17.5)
  Overall fatigue | -6.3 (23.5) | -7.1 (30.8)
  Degree of joint pain | -3.9 (30.2) | -2.3 (24.0)

12. Secondary Outcome: Change From Baseline in Patient and Physician Global Assessments of Disease Activity at Week 24
Description: A participant's overall rating of Disease Activity and a physician's rating of the participant's disease activity. A vertical mark made on a 100 mm line rated 0 (no symptoms) to 100 (severe symptoms) determines the score. Change from baseline was computed as the value at Week 24 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had Patient and Physician Global assessments of Disease Activity at Baseline and Week 24. Data were not available for six participants
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 29 | 17
mm
  Patient Global Assessment of Disease Activity | -14.0 (29.5) | -9.6 (19.1)
  Global Assessment of Disease Activity | -16.4 (16.6) | -13.3 (20.1)

13. Secondary Outcome: Change From Baseline in Patient and Physician Global Assessments of Disease Activity at Week 48
Description: A participant's overall rating of Disease Activity and a physician's rating of the participant's disease activity. A vertical mark made on a 100 mm line rated 0 (no symptoms) to 100 (severe symptoms) determines the score. Change from baseline was computed as the value at Week 48 minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had Patient and Physician Global assessments of Disease Activity at Baseline and Week 48. Data were not available for six participants
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 28 | 18
mm
  Patient Global Assessment of Disease Activity | -9.3 (23.9) | -4.3 (22.0)
  Global Assessment of Disease Activity | -10.1 (22.7) | -8.4 (19.9)

14. Secondary Outcome: Change From Baseline in Tear Secretion as Measured by Schirmer's I Test at Week 24
Description: A paper strip was placed within each lower eyelid and the participant's eyes were closed for 5 minutes. The wet paper was removed after 5 minutes and the length of wetting was recorded to the nearest 0.5 mm. Change from baseline was computed as the value at Week 24 minus the baseline value. A positive value in change from Baseline indicates an improvement and a negative value indicates worsening.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had Schirmer's I test data at Baseline and Week 24. Data were not available for six participants who received baminercept and three participants who received placebo.
Measure: Mean (Standard Deviation); unit: mm/5 min
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 27 | 16
mm/5 min
  Left Eye | 0.8 (8.0) | 1.9 (11.1)
  Right Eye | 1.3 (5.6) | -4.3 (8.5)

15. Secondary Outcome: Change From Baseline in Tear Secretion as Measured by Schirmer's I Test at Week 48
Description: A paper strip was placed within each lower eyelid and the participant's eyes were closed for 5 minutes. The wet paper was removed after 5 minutes and the length of wetting was recorded to the nearest 0.5 mm. Change from baseline was computed as the value at Week 48 minus the baseline value. A positive value in change from Baseline indicates an improvement and a negative value indicates worsening.
Time Frame: Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had Schirmer's I test data at Baseline and Week 48. Data were not available for eight participants who received baminercept and one participant who received placebo.
Measure: Mean (Standard Deviation); unit: mm/5 min
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 25 | 18
mm/5 min
  Left Eye | -0.8 (8.7) | 3.6 (11.2)
  Right Eye | 2.2 (7.4) | 0.2 (9.4)

16. Secondary Outcome: Change From Baseline in Tear Secretion as Measured by Lissamine Green Staining at Week 24
Description: Lissamine green stain was dropped into the participant's eyes and then an ophthalmologist used a slit lamp to examine the eye surface. Six areas of the eye surface were evaluated and scored from 0 to 3, with 0 being no tear film damage to 3, extensive tear film damage. The scores of all six areas in both eyes were totaled to obtain an overall score between 0 and 18. A higher score indicates insufficient tear flow and excessive dryness. Change from baseline was computed as the value at Week 24 minus the baseline value. A negative value in change from Baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had Lissamine Green Staining data at Baseline and Week 24. Data were not available for six participants who received baminercept and three participants who received placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 27 | 16
units on a scale | -0.7 (9.2) | -0.4 (6.3)

17. Secondary Outcome: Change From Baseline in Tear Secretion as Measured by Lissamine Green Staining at Week 48
Description: Lissamine green stain was dropped into the participant's eyes and then an ophthalmologist used a slit lamp to examine the eye surface. Six areas of the eye surface were evaluated and scored from 0 to 3, with 0 being no tear film damage to 3, extensive tear film damage. The scores of all six areas in both eyes were totaled to obtain an overall score between 0 and 18. A higher score indicates insufficient tear flow and excessive dryness. Change from baseline was computed as the value at Week 48 minus the baseline value. A negative value in change from Baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had Lissamine Green Staining data at Baseline and Week 48. Data were not available for eight participants who received baminercept and one participant who received placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 25 | 18
units on a scale | 1.1 (10.8) | 0.1 (9.3)

18. Secondary Outcome: Change From Baseline in the Short Form 36 (SF-36) Physical and Mental Health Component Summary Scores (PCS and MCS) at Week 24
Description: The SF-36 questionnaire completed by the subject measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Summary measures were standardized to have a mean of 50 and a standard deviation of 10 in the 1998 general US population. Change from baseline is computed as the value at Week 24 minus the baseline value. A positive value in change from Baseline indicates an improvement and a negative value indicates worsening.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had SF-36 data at Baseline and Week 24. Data were not available for four participants who received baminercept and two participants who received placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 29 | 17
units on a scale
  Overall Physical Score | 2.7 (6.4) | -1.0 (9.3)
  Overall Mental Score | -1.2 (13.0) | -0.3 (10.3)

19. Secondary Outcome: Change From Baseline in the Short Form 36 (SF-36) Physical and Mental Health Component Summary Scores (PCS and MCS) at Week 48
Description: The SF-36 questionnaire completed by the subject measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Summary measures were standardized to have a mean of 50 and a standard deviation of 10 in the 1998 general US population. Change from baseline is computed as the value at Week 48 minus the baseline value. A positive value in change from Baseline indicates an improvement and a negative value indicates worsening.
Time Frame: Week 48
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either baminercept or placebo and who had SF-36 data at Baseline and Week 48. Data were not available for five participants who received baminercept and one participant who received placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 28 | 18
units on a scale
  Overall Physical Score | 1.4 (6.5) | 1.5 (7.1)
  Overall Mental Score | -1.2 (15.2) | -0.2 (8.3)

20. Secondary Outcome: Percent of Participants With Adverse Events of Grade 3 or Higher
Description: Grades are based on National Cancer Institute--Common Terminology Criteria (NCI-CTCAE) Version 4.0 over the duration of the study. Participants who experienced at least one grade 3 or higher adverse event (AE) are counted only once. The adverse events are treatment-emergent, which means that the AE occurred after taking the first dose of study drug.
Time Frame: From the time of administration of the first dose of study drug until the participant completed study participation, an average of 48 weeks.
Population: The Safety population included all randomized subjects who received at least one dose of either baminercept or placebo.
Measure: Number; unit: Percent of participants
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 33 | 19
Percent of participants | 27.3 | 15.8

21. Secondary Outcome: Percent of Participants With Grade 3 or Higher Infection Adverse Event
Description: Grades are based on National Cancer Institute--Common Terminology Criteria (NCI-CTCAE) Version 4.0 over the duration of the study. Participants who experienced at least one grade 3 or higher infection adverse event (AE) are counted only once. The adverse events are treatment-emergent, which means that the AE occurred after taking the first dose of study drug.
Time Frame: as for outcome 20
Population: The Safety population included all randomized subjects who received at least one dose of either baminercept or placebo.
Measure: Number; unit: Percent of participants
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 33 | 19
Percent of participants | 6.1 | 0

22. Secondary Outcome: Percent of Participants With Injection Site Reaction or Any Grade 2 or Higher Adverse Event Within 24 Hours of Injection
Description: Grades are based on National Cancer Institute--Common Terminology Criteria (NCI-CTCAE) Version 4.0 over the duration of the study. Participants who experienced at least one injection site reaction or Grade 2 or higher adverse event within 24 hours of injection are counted only once. The adverse events are treatment-emergent, which means that the AE occurred after taking the first dose of study drug.
Time Frame: as for outcome 20
Population: The Safety population included all randomized subjects who received at least one dose of either baminercept or placebo.
Measure: Number; unit: Percent of participants
Arm/Group | Baminercept 100 mg | Placebo
Number analyzed (Participants) | 33 | 19
Percent of participants | 81.8 | 57.9

ADVERSE EVENTS:
Time Frame: From the time of administration of the first dose of study drug until the participant completed study participation, an average of 48 weeks.
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (May 28, 2009)
Arm/Group | Baminercept 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/33 | 1/19
Other Adverse Events (participants affected / at risk) | 33/33 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baminercept 100 mg (N=33) | Placebo (N=19)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pleurisy viral (Infections and infestations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baminercept 100 mg (N=33) | Placebo (N=19)
Anaemia (Blood and lymphatic system disorders) | 8 (17) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 8 (11) | 4 (7)
Neutropenia (Blood and lymphatic system disorders) | 4 (7) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 2 (9) | 3 (4)
Injection site haematoma (General disorders) | 3 (3) | 2 (2)
Injection site reaction (General disorders) | 17 (42) | 6 (22)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Vaccination site reaction (General disorders) | 4 (4) | 3 (3)
Hepatobiliary disease (Hepatobiliary disorders) | 2 (2) | 1 (1)
Type IV hypersensitivity reaction (Immune system disorders) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Tooth infection (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (7) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 2 (3)
Blood creatinine increased (Investigations) | 12 (21) | 9 (13)
Weight decreased (Investigations) | 6 (6) | 0 (0)
Weight increased (Investigations) | 4 (4) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 6 (7) | 5 (8)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 (9) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (10) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (3) | 3 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 9 (22) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Randomization was prematurely stopped in July 2014 due to study product expiration. 52 of the 72 planned subjects were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No